CLINICAL TRIAL: NCT00915083
Title: A Phase I Study to Assess the Safety, Pharmacokinetics, and Potential Effects of Amrubicin on the QT/QTc Interval in Cancer Patients With Advanced Solid Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMR PH US 2008 PK002
Record Dates: First submitted 2009-06-04; First posted 2009-06-05 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — amrubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amrubicin 40mg/m^2 (Experimental): Amrubicin 40mg/m^2 given as a 5 minute IV infusion on Days 1, 2 & 3 of a 21 day cycle
  Interventions: Drug: Amrubicin

INTERVENTIONS:
Drug: Amrubicin — 40mg/m^2 5 minute IV infusion for 3 consecutive days (21 day cycle)

SUMMARY:
The purpose of the study is to determine whether amrubicin is safe and effective in the treatment of patients with advanced solid tumors. The study will assess the pharmacokinetics of the amrubicin and if it has an effect on the heart.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting all of the following criteria will be considered for enrollment into the study:

  1. Males or females, aged 18-65 years;
  2. Histological or cytological diagnosis of solid malignancy for which no acceptable standard therapy exists or for which approved standard therapy has failed;
  3. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1;
  4. Life expectancy greater than 3 months;
  5. Nonsmoker or not smoked or used tobacco products for at least 3 months before the screening visit and agree to abstain from smoking/using tobacco products throughout the formal study and until the End of Study visit;
  6. Capable of giving informed consent, has signed the informed consent form, and is willing to comply with scheduled visits, dose administration, and other study procedures;
  7. Women of childbearing potential may participate, providing they have a negative serum pregnancy test (β-HCG) at screening, and a negative urine pregnancy test prior to dosing on Day 1 of each cycle;
  8. Males and females of childbearing potential must agree to the use of at least 2 effective contraceptive methods until at least 28 days following the last dose of study drug;
  9. Serum potassium, magnesium and corrected calcium that is within institutional normal range at screening;
  10. Adequate organ function including the following:

      * Adequate bone marrow reserve: absolute neutrophil count (segmented and bands) (ANC) ≥1.5 x 109/L, platelet count ≥100 x 109/L, and hemoglobin ≥90 g/L,
      * Hepatic: bilirubin ≤1.5 x the upper limit of normal (ULN), ALT and AST ≤2.0 x ULN,
      * Renal: serum creatinine ≤1.5 x ULN or calculated creatinine clearance >80 mL/min.

Exclusion Criteria:

* Patients meeting any of the following criteria will be excluded from the study:

  1. Hypersensitivity to amrubicin or related compounds;
  2. Radiotherapy with curative intent to a primary disease complex ≤ 28 days before first dose; cranial radiotherapy ≤ 21 days before first dose; radiotherapy to all other areas ≤ 7 days before first dose of amrubicin;
  3. History or presence of clinically significant abnormal 12-lead ECG or triplicate ECGs with a mean QT interval corrected for heart rate (HR) using Fridericia's method (QTcF) of >450 msec (males) or >470 msec (females), a PR interval >240 msec or a QRS interval >110 msec (within 3 months of screening visit);
  4. Left ventricular ejection fraction (LVEF) <50%;
  5. Recent history (within 3 months of screening visit) of pericarditis and pericardial effusion;
  6. History within 6 months of the screening visit of one of the following:

     * cardiac disease including congenital long-QT syndrome,
     * angina, congestive heart failure,
     * myocardial ischemia or infarction,
     * myocarditis, chest pain or dyspnea on exertion of cardiac origin,,
     * idiopathic or hypertrophic cardiomyopathy,
     * sarcoidosis,
     * syncope,
     * epilepsy,
     * or other clinically significant cardiac disease;
  7. Family history of long QT syndrome;
  8. Use of implantable pacemaker or implantable cardioverter defibrillator;
  9. Clinically significant bradycardia (<50 beats per minute);
  10. Systolic blood pressure >150 mmHg or diastolic blood pressure >100 mmHg;
  11. Previous treatment with an investigational agent or any anticancer therapy within 4 weeks prior to the 'off-drug' visit;
  12. Previous treatment with anticancer therapy and has not fully recovered (Common Terminology Criteria Adverse Event [CTCAE] Grade 1, except alopecia) from the toxic effects of that treatment;
  13. Treatment with any medication known to produce QT prolongation enzyme-inducing anticonvulsants, non-prescription medications including topical medications, all vitamins, minerals, herbs or dietary supplements/remedies (e.g., Saint John's Wort or Milk Thistle) for at least 7 days before the start of the off-drug visit;
  14. Previous treatment with any anthracycline;
  15. Any condition that would put the patient at undue risk or discomfort as a result of adherence to study procedures;
  16. Women who are pregnant or nursing;
  17. Uncontrolled intercurrent illness such as myelosuppression, renal impairment, hepatic impairment, infection and uncontrolled diabetes;
  18. Symptomatic central nervous system metastases. Patients with asymptomatic brain metastases are allowed. The patient must be stable for ≥ 2 weeks after radiotherapy, if the patient is on corticosteroids, the dose of corticosteroids must have been stable for ≥ 2 weeks prior to the first dose of study treatment, or be in the process of being tapered;
  19. Suspected, diffuse idiopathic interstitial lung disease or pulmonary fibrosis not related to prior treatment;
  20. History of seropositive HIV or patients who are receiving immunosuppressive or myelosuppressive medications that would, in the opinion of the investigator, increase the risk of serious neutropenic complications;
  21. Positive urine drug screen for undeclared concomitant medications and/or illegal drug use at screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-06-01 (Actual); Primary Completion 2011-05-01 (Actual); Study Completion 2011-05-01 (Actual)

PRIMARY OUTCOMES:
To characterize the pharmacokinetics of amrubicin and amrubicinol (metabolite) in plasma, whole blood, and urine in patients given amrubicin as 5 minute IV infusions at 40 mg/m2 for 3 consecutive days; data will be obtained from blood & urine samples | Cycle 1: all primary outcome measures are collected during the first 21 days.
  The duration of making measurements during the first cycle is 21 days. All data relating to the primary outcome measure is collected during this time.
  There is an optional Extension Phase during which subjects can continue to receive additional 21-day cycles of amrubicin unless there is evidence of tumor progression or unacceptable toxicity. The duration of measurements depends on how long the subject continues on treatment.
To evaluate the potential effects on the QT/QTc interval in cancer patients when treated with 5 minute IV infusions of amrubicin 40 mg/m2 daily for 3 consecutive days; data will be obtained by ECG extraction from continuous 12-lead Holter monitoring | Cycle 1: all primary outcome measures are collected during the first 21 days.
  The duration of making measurements during the first cycle is 21 days. All data relating to the primary outcome measure is collected during this time.
  There is an optional Extension Phase during which subjects can continue to receive additional 21-day cycles of amrubicin unless there is evidence of tumor progression or unacceptable toxicity. The duration of measurements depends on how long the subject continues on treatment.
To determine the safety and tolerability of 40 mg/m2 amrubicin given as 5 minute IV infusions for 3 consecutive days; information will be collected by adverse event monitoring and laboratory safety tests. | Cycle 1: all primary outcome measures are collected during the first 21 days.
  The duration of making measurements during the first cycle is 21 days. All data relating to the primary outcome measure is collected during this time.
  There is an optional Extension Phase during which subjects can continue to receive additional 21-day cycles of amrubicin unless there is evidence of tumor progression or unacceptable toxicity. The duration of measurements depends on how long the subject continues on treatment.

SECONDARY OUTCOMES:
1. Explore the relationship between pharmacokinetics and QTc interval change. Information will be obtained by further analysis of the datasets obtained from the primary outcome measures | Cycle 1: all primary outcome measures are collected during the first 21 days.
  The duration of making measurements during the first cycle is 21 days. All data relating to the primary outcome measure is collected during this time.
  There is an optional Extension Phase during which subjects can continue to receive additional 21-day cycles of amrubicin unless there is evidence of tumor progression or unacceptable toxicity. The duration of measurements depends on how long the subject continues on treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Renschler, MD, Study Director — Celgene Corporation
Locations (8):
- United States (8):
  - University of California San Diego, La Jolla, California
  - Sarcoma Oncology Center, Santa Monica, California
  - Indiana University Cancer Pavilion, Indianapolis, Indiana
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Sinai Hospital of Baltimore- Alvin and Lois Lapidus Cancer Institute, Baltimore, Maryland
  - Montefiore Medical Center, The Bronx, New York
  - UT Health Science Center at San Antonio- Cancer Therapy and Research Center, San Antonio, Texas
  - Hunstman Cancer Institute, Salt Lake City, Utah

REFERENCES:
- [Background] Chen N, et al. Phase I study to assess pharmacokinetics (PK), QT/QTc effect, and safety of amrubicin in patients (pts) with advanced solid tumors. Presented at 2011 ASCO Annual Meeting, June 3-7, 2011, Chicaco, IL. Abstract No. 7073 N